CLINICAL TRIAL: NCT05260047
Title: Culturally Responsive Community Driven Substance Use Recovery for Black and Latinx Population
Acronym: IMANI U
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000031168; 1U01OD033241-01 (NIH)
Record Dates: First submitted 2022-02-11; First posted 2022-03-02 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Substance Use; Mental Health Issue; Opioid Use; Medication Assisted Treatment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Referral and Consultation; Genetic Linkage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMANI BREAKTHROUGH (Active Comparator): Participants will participate in 24-week IMANI weekly groups
  Interventions: Behavioral: IMANI
- IMANI BREAKTROUGH + church-based telehealth MAT option (IMANI + CTM) (Experimental): Participants will participate in the 24-week Imani weekly group. During weeks 1-4 participants will received education on MAT. Those participants randomized will receive the IMANI weekly group as well as a church based telehealth Medication Assisted Treatment option. The church based telehealth MAT will consist of participants assigned to receive MAT from addiction treatment providers via telehealth. Telehealth sessions will be provided in the church.
  Interventions: Behavioral: IMANI; Behavioral: Telehealth MAT
- IMANI BREAKTHROUGH + Traditional MAT plus Referral and Linkage (Experimental): Participants will participate in the 24-week Imani weekly group. During weeks 1-4 participants will received education on MAT. Those participants randomized will receive the IMANI weekly group as well as Traditional MAT services with Referral and Linkage to services. Participants in this arm will be provided a list of referrals and links to community MAT providers. They will choose their providers.
  Interventions: Behavioral: IMANI; Behavioral: Traditional MAT plus Referral and Linkage

INTERVENTIONS:
Behavioral: IMANI — For the intervention, the study will introduce and offer Medication Assisted Treatment. Those participants wishing to receive MAT will be randomized to one of two intervention IMANI + church-based telehealth MAT or IMANI + Traditional MAT + Referral and Linkage. Those who do not wish to partake of MAT services will remain in the IMANI alone.
Behavioral: Telehealth MAT — Describe what is the Telehealth MAT briefly
  Arms: IMANI BREAKTROUGH + church-based telehealth MAT option (IMANI + CTM)
Behavioral: Traditional MAT plus Referral and Linkage — Describe what he traditional MAT plus referral and linkage briefly
  Arms: IMANI BREAKTHROUGH + Traditional MAT plus Referral and Linkage

SUMMARY:
The main goal of this current study is to develop and optimize methods for increasing access to, uptake of, and engagement in MAT (Medication Assisted Treatment) among communities of color.

DETAILED DESCRIPTION:
The main goal of this current study is to develop and optimize methods for increasing access to, uptake of, and engagement in MAT (Medication Assisted Treatment) among communities in geographical areas with high overdose cases. Through a multilevel Community Based Participatory Research initiative and a rigorous RCT that incorporates elements of choice in participation, the study will examine whether adding a church-based telehealth MAT option to Imani (Imani + CTM) will improve outcomes for people who reside in geographical areas with high overdose rates with Alcohol Use Disorder or Opioid Use Disorder)compared to Imani + Traditional MAT Referral and Linkage (Imani + Traditional MAT R&L) in the community. Individuals who do not choose to engage in MAT will continue in the Imani group program as usual. Imani (meaning Faith in Swahili) Breakthrough was developed in 2017 through a community based participatory research process. Imani Breakthrough is a faith-based, person-centered, culturally informed harm reduction recovery program that takes place churches in the community in geographical areas with high overdose rates. This program provides an innovative approach to engaging vulnerable groups into Substance Use Disorder treatment by focusing on SAMHSA's 8 dimensions of wellness (social determinants of health), 7 domains of citizenship, culturally informed education, and referral to Medication Assisted Treatment defined as any Food and Drug Administration approved pharmacotherapy for treating Substance Use Disorder. The Community Based Participatory Research process, which incorporates learning from and partnering with the church and larger community (including providers and policymakers), aims to increase the community's understanding of Alcohol Use Disorder and Opioid Use Disorder, tackle Medication Assisted Treatment misconceptions, optimize IMANI implementation, and establish policy recommendations for the healthcare systems to better serve people with Substance Use Disorder.

The specific aims are:

Specific Aim 1: To evaluate the impact of Imani + a church-based telehealth Medicine Assisted Treatment option (Imani + CTM) compared to Imani + Traditional MAT referral and linkage option (Imani + MAT R&L) on medication for addiction treatment initiation and engagement.

Specific Aim 2: To assess whether there are changes in substance use over time for Imani+ CTM compared to Imani + Traditional MAT R&L.

Specific Aim 3: To evaluate potential mediators and moderators (e.g., choice, SDOH) of improvements in primary SUD outcomes (initiation, engagement, and decreased substance use).

Exploratory Aim 1: To assess differences in the 7 domains of citizenship and 8 dimensions of wellness (social determinants of health) comparing those enrolled in a MAT condition to those NOT enrolled in a MAT condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet criteria for a DSM-5 Alcohol Use Disorder and/or Opioid Use Disorder and are currently using alcohol and/or other opioids within the last 28 days.
* Are interested in reducing substance use.
* Self-identify as living in a geographical area with high overdose case rates

Exclusion Criteria:

- Participants who do not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall attendance of program | Up to 24 weeks
  The total number of sessions that participants attend will be used to measure continuation of program.
Overall treatment adherence | Baseline
  The number of participants that adhere to treatments will be measured using self-report at three time points.
Overall treatment adherence | 6-month
  The number of participants that adhere to treatments will be measured using self-report at three time points.
Overall treatment adherence | 12-month
  The number of participants that adhere to treatments will be measured using self-report at three time points.

SECONDARY OUTCOMES:
Change in substance abuse | Weekly for 24 weeks
  Using urine toxicology strips the research staff will test the weekly urine provided by all participants for drugs use.

CONTACTS AND LOCATIONS:
Overall Officials: Chyrell Bellamy, Ph.D., Principal Investigator — Yale University; Ayana Jordan, PhD., Principal Investigator — Yale University
Locations (8):
- United States (8):
  - Mount Aery Baptist Church, Bridgeport, Connecticut
  - Principe of Peace Church, Bridgeport, Connecticut
  - Blackwell Memorial AME Church, Hartford, Connecticut
  - Iglesia Nuevo Comienzo, Hartford, Connecticut
  - Spottswood AME, New Britain, Connecticut
  - Varick Memorial AME Church, New Haven, Connecticut
  - Yale Program for Recovery and Community Health, New Haven, Connecticut
  - Casa de Oracion y Adoracion, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No